CLINICAL TRIAL: NCT04325685
Title: The Effect of Supraglottic and Oropharyngeal Decontamination on the Incidence of Ventilator-associated Pneumonia and Associated Microbiomes.
Brief Title: The Effect of Supraglottic and Oropharyngeal Decontamination on the Incidence of Ventilator-associated Pneumonia
Acronym: SGDC-VAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern State Medical University (Other)
Responsible Party: Principal Investigator, Vsevolod V. Kuzkov, Principal investigator, Northern State Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SGDC-VAP-1
Record Dates: First submitted 2020-03-26; First posted 2020-03-27 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Trauma Injury; Brain Injuries; Abdominal Sepsis; Pancreatitis; Meningitis; Encephalitis; Seizures; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Accidental Injuries; Brain Injuries; Intraabdominal Infections; Pancreatitis; Meningitis; Encephalitis; Seizures; Respiratory Distress Syndrome | interventions — Sodium Chloride; octenidine and phenoxyethanol drug combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator)
  Interventions: Drug: Control
- Antiseptic (Octenisept) group (Active Comparator)
  Interventions: Drug: Antiseptic Solution
- Bacteriophage (Sextaphag) group (Experimental)
  Interventions: Drug: Bacteriophage

INTERVENTIONS:
Drug: Control — Oropharyngeal decontamination with saline will be performing three time a day every 8 hours during mechanical ventilation
  Other Names: Saline
  Arms: Control group
Drug: Antiseptic Solution — Oropharyngeal decontamination with antiseptic solution will be performing three time a day every 8 hours during mechanical ventilation
  Other Names: Octenisept
  Arms: Antiseptic (Octenisept) group
Drug: Bacteriophage — Oropharyngeal decontamination with bacteriophage will be performing three time a day every 8 hours during mechanical ventilation
  Other Names: Sextaphag
  Arms: Bacteriophage (Sextaphag) group

SUMMARY:
Oropharynx is the main source of pathogen microorganisms for the ventilator - associated pneumoniae. As known bacteriophages can eliminate different pathogen microorganisms or reduce a degree of a pathogen's colonization. The research team is considering that oropharyngeal decontamination with bacteriophages can prevent the developing of the ventilator - associated pneumoniae. There will be three groups in this investigation: placebo, antiseptic drug (Octenisept) and bacteriophage (Sexthaphag).

ELIGIBILITY:
Inclusion Criteria:

- invasive mechanical ventilation beyond 48 hours

Exclusion Criteria:

* hospital - acquired pneumonia
* community - acquired pneumoniae
* BMI > 35 kg/cm2
* pregnancy
* tracheostomy
* reintubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
Incidence of ventilator-associated pneumonia (VAP) | Change from Baseline CPIS at 14 days
  CPIS is using for diagnosis the VAP, if CPIS equal or more 6, the VAP will be confirmed
Changing of oral and lung microbiomes | Change from Baseline Microbiology researching at 14 days
  Microbiology researching samples from oral cavity and trachea. The Gram positive and Gram negative aerobes and anaerobes will be assessed with observing Colony Form Unit

SECONDARY OUTCOMES:
Organ dysfunction | Change from Baseline Sequential Organ Function Assessment at 14 days
  Sequential Organ Function Assessment (SOFA) will be using for assessment organ dysfunction Patient examination with Sequential Organ Function Assessment (SOFA). If Sequential Organ Function Assessment more then 2 points Organ dysfunction is present. The hirher value is equal worse outcome
Concentration of C - reactive protein (CRP) | Change from Baseline CRP at 14 days
  Biomarker of the VAP
Concentration of Procalcitonin (PCT) | Change from Baseline PCT at 14 days
  Biomarker of the VAP
Rate of Mortality | Change from Baseline PCT at 28 days
  Mortality for 28 days of a hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Budgetary Healthcare Institution of Arkhangelsk Region "Severodvinsk City Clinical Emergency Hospital # 2", Severodvinsk, Arkhangelskaya oblast, Russia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol